CLINICAL TRIAL: NCT00483925
Title: CARDIOVASCULAR RISK FACTORS IN ADULT PATIENTS WITH MULTISYSTEM LANGERHANS-CELL HISTIOCYTOSIS: EVIDENCE OF GLUCOSE METABOLISM ABNORMALITIES
Brief Title: Cardiovascular Risk Factors and LCH in Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laikο General Hospital, Athens (Other)
Other Study IDs: ES 511
Record Dates: First submitted 2007-06-06; First posted 2007-06-08 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2007-06

CONDITIONS: Histiocytosis, Langerhans-Cell
Keywords: Langerhans cell histiocytosis; flow mediated dilatation; intima media thickness; insulin resistance; hypopituitarism; glucose and lipid metabolism,; structural arterial and functional endothelial properties in patients with multisystem LCH
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell; Insulin Resistance; Hypopituitarism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Langerhans-cell histiocytosis (LCH) is a rare disease with features of chronic inflammation and hypopituitarism, conditions associated with increased risk of cardiovascular diseases.

Objective: To investigate glucose and lipid metabolism, insulin resistance, structural arterial and functional endothelial properties in patients with multisystem LCH in a prospective, observational study.

Interventions:Cardiovascular risk factors: arterial blood pressure, lipid profile, mathematical indices of insulin resistance (IR), intima media thickness, brachial artery flow mediated dilatation, dynamic indices of IR, pituitary function and C-reactive protein will be estimated in patients with LCH and in a control group matched for gender, age, BMI and smoking habits.

DETAILED DESCRIPTION:
CARDIOVASCULAR RISK FACTORS IN ADULT PATIENTS WITH MULTISYSTEM LANGERHANS-CELL HISTIOCYTOSIS: EVIDENCE OF ABNORMALITIES OF CARBOHYDRATE METABOLISM

Langerhans cell histiocytosis (LCH) is a rare disease, usually affecting children although it has recently increasingly been recognized in adults with a prevalence of approximately 1/560.000 cases ( , ). LCH is characterized by the aberrant proliferation of dendritic cells of the monocyte-macrophage system that resemble normal epidermal Langerhans' cells. These cells can infiltrate many sites of the body leading to either localized lesions or widespread systemic disease. Although LCH has been shown to be a clonal disorder ( ) it also exhibits features of an inflammatory disease, as altered expression of cytokines and cellular adhesion molecules important for the migration and homing of Langerhans cell has been documented ( , ). In addition, LCH shows a particular predilection for hypothalamo-pituitary axis (HPA) involvement leading to diabetes insipidus and/ or anterior pituitary dysfunction in 15-50% and 5-20%, of patients respectively (3, , , ). These percentages may be higher in adult patients with multisystem involvement, being 94% and 59% respectively ( ).

The ongoing inflammatory process and the presence of hypopituitarism are considered to be two independent risk factors for cardiovascular diseases probably through the induction of insulin resistance (IR) ( , , ). The various therapies used for the treatment of multisystem LCH, chemotherapy, radiotherapy and particularly glucocorticoids, may also adversely affect the cardiovascular system mostly through IR ( , ). It is therefore possible that patients with LCH represent a group at higher risk for cardiovascular diseases through the additive effect of a number of different contributing mechanisms known to induce IR. Insulin resistance besides producing an adverse metabolic profile can also lead to endothelial dysfunction and early vascular disease ( ). Early vascular disease can be detected by non-invasive surrogate markers, such as intima-media thickness (IMT) for vascular structure properties and flow-mediated vasodilatation (FMD) for vascular functional properties ( , , ). Carotid IMT is considered an established marker for early atherosclerotic disease and predictor of future cardiovascular events (16) whereas brachial artery FMD has been correlated with coronary endothelial function, a well-known predictor of future cardiovascular events (18).

Main outcome measures: Cardiovascular risk factors assessment were estimated in patients with LCH and compared to controls; the effect of hypopituitarism, disease activity and/ or treatment were determined.

SUBJECTS AND METHODS All patients have to fulfil the diagnostic criteria for "definitive diagnosis" of LCH ( ). Matched to sex, age, and BMI healthy individuals, in good health and not receiving any medication known to affect carbohydrate, sex hormone metabolism, and/or endothelial function for at least 3 months prior have also to be recruited for the study.

Clinical data of the patients as well as hormonal and imaging assessment will be registered.

All subjects do not have participate in strenuous physical activities and have to be on a balanced isocaloric diet for at least 4 weeks prior to the study. Current smokers will be asked not to smoke one day before the hemodynamic study.

Cardiovascular risk factors assessment:

Clinical cardiovascular risk:

* BMI
* waist circumference
* systolic (SBP) and diastolic (DBP) blood pressure Metabolic Profile

The metabolic study of all patients will be performed after a 10h overnight fasting:

* Oral glucose tolerance test
* Glucose, insulin
* Total cholesterol, HDL-cholesterol, triglycerides
* Indices of Insulin resistance [GIR ( ), HOMA ( ), QUICKI ( ), MATSUDA ( ), glucose and insulin response to glucose by calculating the area under the curve (AUC) during the OGTT performance for glucose (AUCGLU) and insulin (AUCINS), using the trapezoidal rule, predicted index of first phase of insulin secretion, predicted index of second phase of insulin secretion ( )].

Hemodynamic studies

* The hemodynamic study will be performed, the day after the metabolic study. Both functional and structural arterial properties will be assessed by non-invasive, easily reproducible hemodynamic ultrasonographic methods, namely: IMT measurement in carotid arteries and both endothelium-dependent FMD and endothelium-independent nitrate-induced dilatation (NID) measurement in brachial artery. IMT, FMD and NID were measured by B-Mode high-resolution ultrasound imaging (VIVID PRO; GENERAL ELECTRIC) ( ).
* Arterial stiffness will be assessed by Applanation Tonometry (SphygmocorTM PWV MEDICAL) on radial artery.

Inflammatory index C-reactive protein (CRP) measurement. References Baumgartner I, von Hochstetter A, Baumert B, Luetolf U, Follath F 1997 Med Pediatr Oncol 28:9-14

* Dunger DB, Broadbent V, Yeoman E, Seckl JR, Lightman SL, Grant DB, Pritchard J 1989 The frequency and natural history of diabetes insipidus in children with Langerhans-cell histiocytosis N Engl J Med 321:1157-1162
* Willman CL, Busque L, Griffith BB, Favara BE, McClain KL, Duncan MH, Gilliland DG 1994 Langerhans'-cell histiocytosis (histiocytosis X)--a clonal proliferative disease N Engl J Med 331:154-160
* de Graaf JH, Tamminga RY, Dam-Meiring A, Kamps WA, Timens W 1996 The presence of cytokines in Langerhans' cell histiocytosis J Pathol 180:400-40
* Egeler RM, Favara BE, van Meurs M, Laman JD, Claassen E 1999 Differential In situ cytokine profiles of Langerhans-like cells and T cells in Langerhans cell histiocytosis: abundant expression of cytokines relevant to disease and treatment Blood 94:4195-4201
* Malpas JS 1998 Langerhans cell histiocytosis in adults Hematol Oncol Clin North Am 12:259-26
* Willis B, Ablin A, Weinberg V, Zoger S, Wara WM, Matthay KK 1996 Disease course and late sequelae of Langerhans' cell histiocytosis: 25-year experience at the University of California, San Francisco J Clin Oncol 14:2073-2082
* Grois NG, Favara BE, Mostbeck GH, Prayer D 1998 Central nervous system disease in Langerhans cell histiocytosis Hematol Oncol Clin North Am 12:287-305
* Makras P, Samara C, Antoniou M, Zetos A, Papadogias D, Nikolakopoulou Z, Andreakos E, Toloumis G, Kontogeorgos G, Piaditis G, Kaltsas GA 2006 Evolving radiological features of hypothalamo-pituitary lesions in adult patients with Langerhans cell histiocytosis (LCH) Neuroradiology 48:37-44
* Alexander RW 1994 Inflammation and coronary artery disease N Engl J Med. 1994 Aug 18;331(7):468-9
* Rosen T, Bengtsson BA 1990 Premature mortality due to cardiovascular disease in hypopituitarism Lancet 336:285-288
* Wilson PW, Kannel WB, Silbershatz H, D'Agostino RB 1999 Clustering of metabolic factors and coronary heart disease Arch Intern Med 159:1104-1109
* Wei L, MacDonald TM, Walker BR 2004 Taking glucocorticoids by prescription is associated with subsequent cardiovascular disease Ann Intern Med 141:764-770
* Andrews RC, Walker BR 1999 Glucocorticoids and insulin resistance: old hormones, new targets. Clin Sci (Lond) 96:513-523

W Wheatcroft SB, Williams IL, Shah AM, Kearney MT 2003 Pathophysiological implications of insulin resistance on vascular endothelial function Diabet Med 20:255-268

Hodis HN, Mack WJ, LaBree L, Selzer RH, Liu CR, Liu CH, Azen SP 1998 The role of carotid arterial intima-media thickness in predicting clinical coronary events.

Ann Intern Med 128:262-269

Schachinger V, Britten MB, Zeiher AM 2000 Prognostic impact of coronary vasodilator dysfunction on adverse long-term outcome of coronary heart disease.

Circulation 101:1899-1906

Anderson TJ, Uehata A, Gerhard MD, Meredith IT, Knab S, Delagrange D, Lieberman EH, Ganz P, Creager MA, Yeung AC, et al 1995 Close relation of endothelial function in the human coronary and peripheral circulations J Am Coll Cardiol 26:1235-1241

Arico M, Girschikofsky M, Genereau T, Klersy C, McClain K, Grois N, Emile JF, Lukina E, De Juli E, Danesino C 2003 Langerhans cell histiocytosis in adults. Report from the International Registry of the Histiocyte Society Eur J Cancer 39:2341-2348

Legro RS, Finegood D, Dunaif A 1998 A fasting glucose to insulin ratio is a useful measure of insulin sensitivity in women with polycystic ovary syndrome J Clin Endocrinol Metab 83:2694-2698

Bergman RN, Prager R, Volund A, Olefsky JM 1987 Equivalence of the insulin sensitivity index in man derived by the minimal model method and the euglycemic glucose clamp J Clin Invest 79:790-800

Katz A, Nambi SS, Mather K, Baron AD, Follmann DA, Sullivan G, Quon MJ 2000 Quantitative insulin sensitivity check index: a simple, accurate method for assessing insulin sensitivity in humans J Clin Endocrinol Metab 85:2402-2410

Matsuda M, DeFronzo RA 1999 Insulin sensitivity indices obtained from oral glucose tolerance testing. Comparison with the euglycemic insulin clamp Diabetes Care 22:1462-1470

Stumvoll M, Mitrakou A, Pimenta W, Jenssen T, Yki-Jarvinen H, Van Haeften T, Renn W, Gerich J Use of the oral glucose tolerance test to assess insulin release and insulin sensitivity Diabetes Care 295-301

Alexandraki K, Protogerou A, Papaioannou TG, Piperi C, Mastorakos G, Lekakis J, Panidis D, Diamanti-Kandarakis E 2006 Early Microvascular and Macrovascular Dysfunction is not Accompanied by Structural Injury in Polycystic Ovary Syndrome. HORMONES (Athens Greece) 5:126-136

ELIGIBILITY:
Inclusion Criteria:

* diagnostic criteria for "definitive diagnosis" of LCH

Exclusion Criteria:

* not participate in strenuous physical activities, on a balanced isocaloric diet for at least 4 weeks prior to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2005-09

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Kaltsas, MD, FRCP, Study Director — Division of Endocrinology, Department of Pathophysiology, Laiko University Hospital
Locations (1):
- Division of Endocrinology, Department of Pathophysiology, Laiko University Hospital,, Athens, Greece

REFERENCES:
- [Background] Alexandraki K, Protogerou AD, Papaioannou TG, Piperi C, Mastorakos G, Lekakis J, Panidis D, Diamanti-Kandarakis E. Early microvascular and macrovascular dysfunction is not accompanied by structural arterial injury in polycystic ovary syndrome. Hormones (Athens). 2006 Apr-Jun;5(2):126-36. doi: 10.14310/horm.2002.11176. PMID 16807225
- [Background] Makras P, Samara C, Antoniou M, Zetos A, Papadogias D, Nikolakopoulou Z, Andreakos E, Toloumis G, Kontogeorgos G, Piaditis G, Kaltsas GA. Evolving radiological features of hypothalamo-pituitary lesions in adult patients with Langerhans cell histiocytosis (LCH). Neuroradiology. 2006 Jan;48(1):37-44. doi: 10.1007/s00234-005-0011-x. Epub 2005 Nov 15. PMID 16292545
- [Result] Arico M, Girschikofsky M, Genereau T, Klersy C, McClain K, Grois N, Emile JF, Lukina E, De Juli E, Danesino C. Langerhans cell histiocytosis in adults. Report from the International Registry of the Histiocyte Society. Eur J Cancer. 2003 Nov;39(16):2341-8. doi: 10.1016/s0959-8049(03)00672-5. PMID 14556926